CLINICAL TRIAL: NCT03092804
Title: The Brain Structure and Neural Network Changing the Before and After Ventriculo-peritoneal Shunting in the Normal Pressure Hydrocephalus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroimagingNPH
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Shunting; Brain constructure; Neural network
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- normal pressure hydrocephalus: Included will be subjects with a probable diagnosis of NPH. The diagnosis will be based primarily on presence of gait impairment plus at least one other impairment in urinary symptoms, cognition impairment or both
  The NPH patients will undergo the CSF tap test and then receive the ventriculo-peritoneal shunting surgery. They will have the examination of brain constructure neuroimaging and functional MRI prior to and posterior to the shunting.
  Interventions: Procedure: ventriculo-peritoneal shunting
- normal control: Healthy volunteers will undergo the examination of brain constructure and functional MRI.

INTERVENTIONS:
Procedure: ventriculo-peritoneal shunting — A mainstream therapy for NPH. It involves the device of CSF flow control of shunts and accessories(CFDA(I)20143665605)
  Groups: normal pressure hydrocephalus

SUMMARY:
With the advent of the aging society, dementia becomes the focus of common people. As for the neurodegeneration dementia, no disease modifying treatments have been discovered. Idiopathic normal pressure hydrocephalus (iNPH) is considered as one of reversible dementia, which can be hint by the surgery. In addition, dementia of iNPH is the typical subcortical dementia. Therefore exploring the pathogenic mechanism is conducive to the early diagnosis and treatment. This research is to monitor the changing of iNPHGS, cognitive function, walking ability as well as brain construction imaging and neural network before and after ventriculo-peritoneal shunting in order to demonstrate the pathogenesis of triads. In the process, the supplementary test, for instance, CSF tap test, will be validated the predictive value.

ELIGIBILITY:
Inclusion Criteria:

ncluded will be subjects with a probable diagnosis of NPH. The diagnosis will be based primarily on presence of gait impairment plus at least one other impairment in urinary symptoms, cognition impairment or both.

1. Are 50 years old or older
2. Patients who understand the study protocol
3. Patients who meet the criteria for NPH

   1. A typical personal history
   2. A typical brain imaging on head CT or MRI
   3. Normal LP findings excluding other conditions
   4. Exclusion of other conditions causing the symptomatology

Exclusion Criteria:

1. Patients below the age of 50 years.
2. Patients who underwent shunt surgery before

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with physical and cognitive symptoms and brain image ﬁndings (Brain CT or MRI) suggestive of NPH were evaluated at neurological outpatient clinic of Peking Union Medical College Hospital according to the NPH diagnosis criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
The brain constructure and neural network changing one day after shunting | Day 1 after shunting
  * Using the voxel based morphology technique to measure the ventricular volume and brain lobe volume
  * Neural network( DMN)by the resting functional MRI
The brain constructure and neural network changing 90 days after shunting | Day 90 after shunting
  Using the voxel based morphology technique to measure the ventricular volume and brain lobe volume
  •Neural network( DMN)by the resting functional MRI
The brain constructure and neural network changing one year after shunting | one year after shunting
  Using the voxel based morphology technique to measure the ventricular volume and brain lobe volume
  •Neural network( DMN)by the resting functional MRI

SECONDARY OUTCOMES:
Assessment of the clinical syndrome of normal pressure hydrocephalus | Day 1 after shunting
  iNPHGS
Assessment of the clinical syndrome of normal pressure hydrocephalus | Day 90 after shunting
  iNPHGS
Assessment of the clinical syndrome of normal pressure hydrocephalus | one year after shunting
  iNPHGS

OTHER OUTCOMES:
Cognition assessments | Day 1 after shunting
  The neuropsychological battery assessment (including MMSE, MOCA as well as cognitive domains especially executive function examinations)
Cognition assessments | Day 90 after shunting
  The neuropsychological battery assessment (including MMSE, MOCA as well as cognitive domains especially executive function examinations)
Cognition assessments | one year after shunting
  The neuropsychological battery assessment (including MMSE, MOCA as well as cognitive domains especially executive function examinations)
Walking ability evaluation | Day 1 after shunting
  Including 10m walking test, up and go tests
Walking ability evaluation | Day 90 after shunting
  Including 10m walking test, up and go tests
Walking ability evaluation | one year after shunting
  Including 10m walking test, up and go tests

CONTACTS AND LOCATIONS:
Overall Officials: Jing Gao, MD, Principal Investigator — Department of Neurology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No